CLINICAL TRIAL: NCT06080763
Title: Exploring Biomechanics and Clinical Outcomes in Responders and Non-Responders to Physical Therapy Management for Knee Osteoarthritis
Brief Title: Biomechanics and Clinical Outcomes in Responders and Non-Responders
Status: Recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Komsak Sinsurin, Asst.Prof.Dr. Komsak Sinsurin, Mahidol University
Other Study IDs: MU-CIRB 2023/117.1108
Record Dates: First submitted 2023-09-22; First posted 2023-10-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis, Knee; Arthroplasty, Replacement, Knee; Physical Therapy
Keywords: Biomechanics; Assessment, Outcomes
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Responders: Individuals who do not respond to physical therapy are determined by the absence of significant improvements, with no change in pain or function exceeding 50%, and with an absolute change of less than 20%.
  Interventions: Procedure: Physical Therapy Management
- Responders: Individuals who respond to physical therapy are determined by the presence of significant improvements, with changes in pain or function exceeding 50%, and with an absolute change of more than 20%.
  Interventions: Procedure: Physical Therapy Management

INTERVENTIONS:
Procedure: Physical Therapy Management — Physical therapy management is a routine intervention provided by physical therapists at Mahidol University's Physical Therapy Center for individuals with knee osteoarthritis.

SUMMARY:
Knee osteoarthritis is a degenerative joint disease that affects many older adults. However, not all patients see improvements as a result of physical therapy management; therefore, a better understanding of biomechanics and assessment of clinical outcomes between responders and non-responders is required.

The included participants will be provided with informed consent and an explanation of the study procedure before enrolling in data collection. The data collection will be arranged in the same order. Practice trials will be provided before the start of data collection. The data collection will consist of standardized questionnaires, assessments, and tests commonly used in clinics.

DETAILED DESCRIPTION:
During data collection, markerless motion capture systems will be placed around the area of interest. The markerless system does not require markers to be attached to the participant's body.

The data collection will include:

1. Demographic information such as age, sex, body height, body weight, body mass index, medical history, medical diagnosis, and the Kellgren-Lawrence score.
2. Patient-reported questionnaires such as the numeric pain rating scale, knee injury and osteoarthritis outcome score, Western Ontario and McMaster Universities Osteoarthritis, and Depression, Anxiety, and Stress Scale - 21 Items.
3. Clinical assessments such as the Varus-valgus laxity test, Foot posture index, Range of motion, Muscle flexibility, and Muscle strength.
4. Functional tests such as the Timed up and go test, Five times sit-to-stand test, Four-meter walk test, and Bipedal quiet stance test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee osteoarthritis based on American College of Rheumatology
* Pain intensity of ≥ 4 out of 10 at the pre-treatment day
* Ability to walk for at least six meters without an assistive device

Exclusion Criteria:

* History of previous lower limb surgery, such as total hip replacement
* History of neurological disorder, such as stroke
* History of vestibular disease, such as Meniere's disease

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with knee osteoarthritis who are currently receiving physical therapy management at Mahidol University's Physical Therapy Center
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Pain intensity will be measured at four time points (i.e., pre-treatment, 6-sessions treatment, 12-sessions treatment, and 18-sessions treatment) spanning up to 6 months.
  The pain intensity will be measured using a numeric rating scale from 0 to 10, with 0 indicating no pain and 10 representing the worst pain imaginable.
Knee Injury and Osteoarthritis Outcome Score | Knee injury and osteoarthritis outcome score will be measured at four time points (i.e., pre-treatment, 6-sessions treatment, 12-sessions treatment, and 18-sessions treatment) spanning up to 6 months.
  The Knee Injury and Osteoarthritis Outcome Score is a questionnaire designed to assess participants' perceptions of their knee severity in various contexts. This questionnaire comprises 42 items that evaluate the participant's perception of pain, stiffness, function, and other knee-related symptoms. Each item is rated on a five-point Likert scale, with 0 indicating no problem and 4 indicating extreme problems. The total score will be transformed to range from 0 to 100 percent.
Western Ontario and McMaster Universities Osteoarthritis | Western Ontario and McMaster Universities Osteoarthritis will be measured at four time points (i.e., pre-treatment, 6-sessions treatment, 12-sessions treatment, and 18-sessions treatment) spanning up to 6 months.
  The Western Ontario and McMaster Universities Osteoarthritis is a questionnaire to assesses the level of pain, stiffness, and physical functioning in individuals with knee osteoarthritis. The questionnaire consists of 24 items that are divided into three subscales: 1) pain (5 items); 2) stiffness (2 items); and 3) physical function (17 items). Each item is rated on a five-point Likert scale, with 0 indicating no pain or difficulty and 4 indicating extreme pain or difficulty. The scores for each subscale are summed up, with a possible score range of 0-20 for pain, 0-8 for stiffness, and 0-68 for physical function.
Depression, Anxiety and Stress Scale - 21 Items | Depression, Anxiety and Stress Scale - 21 Items will be measured at four time points (i.e., pre-treatment, 6-sessions treatment, 12-sessions treatment, and 18-sessions treatment) spanning up to 6 months.
  The Depression, Anxiety and Stress Scale - 21 Items is a self-report questionnaire designed to measure the severity of symptoms related to depression, anxiety, and stress. It consists of 21 items, with seven items dedicated to each of the three domains: 1) depression (7 items); 2) anxiety (7 items); and 3) stress (7 items). Each item is scored on a four-point Likert scale, with 0 indicating that the symptom is not present and 3 indicating that the symptom is severe. The scores for each domain are summed and then multiplied by two, resulting in a possible score range of 0-42 for depression, 0-42 for anxiety, and 0-42 for stress.
Varus-valgus laxity score | Varus-valgus laxity score will be measured at four time points (i.e., pre-treatment, 6-sessions treatment, 12-sessions treatment, and 18-sessions treatment) spanning up to 6 months.
  The varus-valgus laxity test is an assessment used to evaluate the stability of the knee joint. Laxity will be graded based on the amount of medial movement observed: 0 for no movement, 1 for slight medial movement of 5-10 mm, and 2 for substantial medial movement greater than 10 mm. The score will range from 0 to 2.
Foot posture index | Foot posture index will be measured at four time points (i.e., pre-treatment, 6-sessions treatment, 12-sessions treatment, and 18-sessions treatment) spanning up to 6 months.
  The foot posture index is an assessment used to evaluate the posture of the foot and identify any deviations from normal alignment. The foot posture index involves the evaluation of six different aspects of foot posture: 1) talar head palpation; 2) supra and inferolateral malleolar curvature; 3) calcaneal eversion/inversion; 4) bulge in the region of the talonavicular joint; 5) height and congruence of the medial longitudinal arch; and 6) abduction/adduction of the forefoot. Each aspect is scored on a scale ranging from -2 to +2, with 0 representing a neutral or "normal" position. The final score ranges from -12 to +12. A more negative number indicates a supinated foot, while a more positive number indicates a pronated foot.
Muscle flexibility | Muscle flexibility will be measured at four time points (i.e., pre-treatment, 6-sessions treatment, 12-sessions treatment, and 18-sessions treatment) spanning up to 6 months.
  The muscle flexibility is used to evaluate the ability of muscles to lengthen. The flexibility of the quadriceps, hamstring, and gastrocnemius will be measured. The results will be reported in degrees.
Range of motion | Range of motion will be measured at four time points (i.e., pre-treatment, 6-sessions treatment, 12-sessions treatment, and 18-sessions treatment) spanning up to 6 months.
  Range of motion is used to evaluate joint mobility during active movement. The range of motion for the hip, knee, and ankle joints will be measured. The results will be reported in degrees.
Muscle strength | Muscle strength will be measured at four time points (i.e., pre-treatment, 6-sessions treatment, 12-sessions treatment, and 18-sessions treatment) spanning up to 6 months.
  Muscle strength is used to evaluate the maximum force generated by muscles. The strength of the hip extensor, hip abductor, and knee extensor will be measured. The results will be reported in newtons.
Joint kinematics | Joint kinematics will be measured at four time points (i.e., pre-treatment, 6-sessions treatment, 12-sessions treatment, and 18-sessions treatment) spanning up to 6 months.
  Joint kinematics is used to evaluate the movement of the trunk, hip, and knee joints during functional tests such as the Timed Up and Go Test, Five Times Sit-to-Stand Test, Four-Meter Walk Test, and Bipedal Quiet Stance Test. The results will be reported in degrees per second.

CONTACTS AND LOCATIONS:
Overall Officials: Komsak Sinsurin, Ph.D., Principal Investigator — Biomechanics and Sports Research unit, Faculty of Physical Therapy, Mahidol University; Phunsuk Kantha, Ph.D., Principal Investigator — Faculty of Physical Therapy, Mahidol University
Locations (2):
- Thailand (2):
  - Physical Therapy Center, Mahidol University, Bangkok, Bang Phlat
  - Faculty of Physical Therapy, Mahidol University, Nakhon Pathom, Salaya

IPD SHARING:
Plan to Share IPD: Undecided